CLINICAL TRIAL: NCT06897956
Title: Effect of Oral Health Educational Program on Oral Hygiene Knowledge and Practices in a Group of Orphan Children: A Before and After Study
Brief Title: Oral Health Educational Program on Oral Hygiene Knowledge and Practices in a Group of Orphan Children
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Abdelgawad, Associate Professor, Cairo University
Other Study IDs: CEBD-CU-2025-02-13
Record Dates: First submitted 2025-02-13; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Dental Caries; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Dental Caries; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Wadi Hof Orphanage children: Orphan children at that Wadi Hof Branch
  Interventions: Other: Oral health educational program
- El-Doki Orphanage children: Orphan children at that El-Doki Branch
  Interventions: Other: Oral health educational program
- Helwan Orphanage children: Orphan children at that Helwan Branch
  Interventions: Other: Oral health educational program
- Misr Elgadida Orphanage children: Orphan children at that Misr Elgadida Branch
  Interventions: Other: Oral health educational program
- 6th October Orphanage children: Orphan children at that 6th October Branch
  Interventions: Other: Oral health educational program

INTERVENTIONS:
Other: Oral health educational program — Oral health educational program about oral hygiene, prevention of dental caries and techniques of tooth brushing

SUMMARY:
An orphan is defined as "a child under the age of 18 whose mother, father, both parents, and a primary caregiver has died, and who is in need of care or protection". Orphans, therefore, are considered disadvantaged and socially marginalized population whom diseases burden is high. Egypt has 1.7 million orphaned children. The number of children between the age of 0 and 17 who are currently registered in orphanages is 12,015. Dental diseases especially plaque, gingival and dental caries are highly preventable, with the highest prevalence in the developing countries. Profound disparities exist in oral health status across different social and economic divisions. The pattern of orphanage living is quite different from family living as the latter provides physical security, food, and shelter but is devoid of psychological security. High prevalence of dental caries, gingivitis and dental trauma has been observed in children of orphanages. This has been attributed to many factors such as: lack of adequate staff, poor oral hygiene, improper nutrition and eating patterns, high consumption of sugary food, negligence of tooth brushing, moreover the children and caregivers knowledge, level of education and oral health illiteracy. Untreated oral diseases could lead to psychological and general health problems, pain and loss in school time. Recognition of these problems is essential to provide optimum oral health for these deprived children. Health education is an important tool of public health and an effective primary preventive method especially for school aged children in controlling plaque, gingival and dental diseases.

DETAILED DESCRIPTION:
The aim of this study is to raise more awareness about the causes of dental diseases (plaque, gingival and dental caries and their prevention through implementing an educational program to the orphan children focusing on tooth brushing, proper use of fluoride products and proper nutrition. The objectives of this study are to evaluate the impact of the oral health education program on the Knowledge and practices of the orphans and also its effect on the gingival health and dental caries among the children in different branches of orphanages in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Orphan Children aged 7 years old and above.
* Educated children.
* No learning difficulty.
* No medical conditions.

Exclusion Criteria:

* Any child that refuses to participate

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study is carried out at orphanages from different branches in Egypt. The study was conducted using a convenient sample of orphan children aged 7years and above.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Oral hygiene knowledge, and practices of the orphan children | Before the educational program and after 2 months
  Questionnaire including 20 questions about the oral hygiene knowledge and practices of the children. This questionnaire was used before the educational program and after 2 months from the program

SECONDARY OUTCOMES:
Dental Caries experience for permanent dentition | Before the educational program and after 2 months
  DMF index for permanent teeth
Dental Caries experience for mixed dentition | Before the educational program and after 2 months
  Both dental caries indices (DMF and def) are used to provide the caries experience of each participant, they are not added together and reported separately as mixed dentition has both primary and permanent teeth, so we need to record primary teeth with def and permanent teeth with DMF
Oral hygiene | Before the educational program and after 2 months
  Oral Hygiene Index-Simplified which is assessed through scores from 0-3

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided